CLINICAL TRIAL: NCT04251741
Title: Using Adalimumab Serum Concentration to Choose a Subsequent Biological DMARD in Rheumatoid Arthritis Patients Failing Adalimumab Treatment: a Blinded Randomized Superiority Trial
Brief Title: Using Adalimumab Serum Concentration to Choose a Subsequent Biological DMARD in Rheumatoid Arthritis Patients Failing Adalimumab Treatment
Acronym: ADDORA-switch
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Reade Rheumatology Research Institute (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADDORA-switch
Record Dates: First submitted 2020-01-08; First posted 2020-02-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Adalimumab; Rheumatoid arthritis; Therapeutic Drug Monitoring; Drug level; Switching; Failure; Non-response; Subsequent biological
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Patients with rheumatoid arthritis starting another bDMARD after adalimumab failure (defined as DAS28CRP>2.9) are randomly assigned to usual care (with randomized switch to etanercept or to a non-TNF-inhibitor) or 'drug concentration' guided switch.
  When randomized to the usual care group, the treating rheumatologist gets the advice from an independent coworker to switch patients to etanercept 1*50 mg/week or a non-TNFi (abatacept, rituximab, tocilizumab, or sarilumab), based on random allocation. When randomized to a non-TNFi, the treating rheumatologist will choose the non-TNFi. In the 'drug concentration guided' group, in patients with a concentration <1.0 mg/L a switch to etanercept (standard dosing regimen of 50mg once a week) is advised by an independent coworker and in patients with a concentration ≥ 1.0 start of a non-TNF-inhibitor (the same drugs and dosing as in usual care group) is advised.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Rheumatologists and patients remain blinded for allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care group (Active Comparator): Based on a secondary randomization schedule patients are treated with etanercept or a non-TNFi (abatacept, rituximab, tocilizumab, or sarilumab)
  Interventions: Other: Usual care
- 'Drug concentration guided' group (Experimental): Patients with a concentration <1.0 mg/L switch to etanercept and patients with a concentration ≥ 1.0 start a non-TNFi (abatacept, rituximab, tocilizumab, or sarilumab)
  Interventions: Diagnostic Test: Adalimumab trough concentration

INTERVENTIONS:
Diagnostic Test: Adalimumab trough concentration — In the 'drug concentration guided' group, switching to subsequent biological is based on adalimumab trough concentration
  Arms: 'Drug concentration guided' group
Other: Usual care — In the usual care group, switch to subsequent biological is based on secondary randomisation
  Arms: Usual care group

SUMMARY:
A potential application of therapeutic drug monitoring is to predict efficacy after switch to another biological in the case of inefficacy of the previous TNF-inhibitor (TNFi) in rheumatoid arthritis (RA) patients. It has been shown that when antidrug antibodies against adalimumab are detected (resulting in lower drug serum concentrations) in patients failing adalimumab, a normal response to a next TNF blocker can be anticipated. However, when clinical response is unsatisfactory and no antidrug antibodies against the first TNFi are detected (generally drug levels are adequate in this case), this predicts a lower response to a next TNFi. This means drug resistant failure in the former, compared to class resistant failure in latter category of patients. The current RA treatment strategy after failure of the first TNF-inhibitor is to start either a second TNFi or a non-TNFi. However, by channelling patients with sufficient adalimumab concentration to a non-TNFi will provide higher chance of disease control. Patients with very low or undetectable drug levels have an equal or potential higher chance of disease control with a drug of the same class (i.e. another TNFi).

DETAILED DESCRIPTION:
Over the last decades biopharmaceuticals such as agents against tumor necrosis factor (TNF), are frequently prescribed to optimize rheumatoid arthritis treatment. Although TNFi such as adalimumab, etanercept and infliximab, have improved the treatment of rheumatoid arthritis, a proportion of patients discontinue the treatment because of inefficacy or intolerance.

Where TNFi have failed, mainly two treatment approaches are available: switch to another TNFi or to a biological with a different mode of action (notably rituximab, abatacept or tocilizumab) or to a target synthetic DMARDs. The EULAR recommendation for the management of rheumatoid arthritis advocate that any biologic agent including a subsequent TNFi can be used with equal chance for effect in case of non-response to a previous TNFi. This recommendation is based on three randomized controlled trails, but it should be noted that systematic reviews also including non-randomized controlled studies sometimes concluded that non-TNFi are more effective after TNFi failure than a second TNFi.

Of note, currently there are no strong predictors available for response to bDMARDS in RA. This study focuses on non-response after adalimumab, as this is the most prescribed TNFi worldwide.

Although it seems that indeed on a group level response to a non-TNFi is comparable to a second TNFi after the first TNFi has failed, using therapeutic drug monitoring could identify subgroups of patient who would benefit more from either a non-TNFi or a TNF-i as next treatment. The underlying pathophysiological mechanisms for this hypothesis are explored in this study.

Nonresponse on adalimumab in RA can have different causes. Firstly, the patient might not be sensitive to TNF blockade at all, or the patient develops this trait later on (primary nonresponse or secondary nonresponse). In these patients, switching to a non-TNFi might conceptually be superior to starting a second TNFi. However, in other patients nonresponse (either primary or secondary) might be caused by inefficient drug concentration because of development of antidrug antibodies against adalimumab. In these patients a TNFi might be just as effective as a non-TNFi, as these patients have drug- but not class failure. Thus, testing of adalimumab levels might be helpful in channelling patients to their most optimal treatment.

Above mentioned hypothesis has been tested in three studies (5) of which one concerned adalimumab in RA. This study showed that response to a second TNFi was indeed higher in patients with antidrug antibodies (ADA) and low adalimumab levels, and lower in patients with adequate adalimumab levels. However, a diagnostic study comparing a serum concentration guided versus usual care switching strategy has not yet been performed.

In this multi-centre, double blinded randomized controlled trial it will be evaluated whether clinical outcome after switching to a subsequent biological treatment is superior with a switching strategy using adalimumab concentration compared to usual care switching strategy.

Patients with rheumatoid arthritis starting another bDMARD (biologic disease modifying antirheumatic drugs) after adalimumab failure (defined as DAS28-CRP >2.9) are randomly assigned to usual care (with randomized switch to etanercept or to a non-TNFi) or 'drug concentration' guided switch.

Data regarding disease status, functioning, adverse events and use of co-medication/rescue medication will be collected during this study.

ELIGIBILITY:
Inclusion Criteria:

* rheumatoid arthritis patient, according to American College of Rheumatology (ACR) 1987 and/or EULAR/ACR 2010 criteria;
* recently failed treatment with adalimumab (defined as DAS28-CRP >2.9) and not treated with a subsequent bDMARD or target synthetic DMARD (tsDMARD)
* Received adalimumab for at least 10 weeks in standard dosing (40mg subcutaneously every other week, either in monotherapy or combined with methotrexate or leflunomide)
* Stop adalimumab due to inefficacy, either alone or combined with side effects
* who has agreed to participate (written informed consent);
* age 16 years or older.

Exclusion Criteria:

* Treatment with another TNF-inhibitor prior to adalimumab
* Treatment with all non-TNFi options (abatacept, rituximab, sarilumab and tocilizumab) prior to adalimumab
* scheduled surgery during the follow-up of the study or other pre-planned reasons for treatment discontinuation
* life expectancy shorter than follow-up period of the study;
* no possibility to safely receive an TNF-inhibitor or a non TNF-inhibitor

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
mean time weighted DAS28-CRP | 24 weeks
  difference in mean time weighted DAS28-CRP between the two groups

SECONDARY OUTCOMES:
Good or moderate response according the EULAR response criteria | 12 en 24 weeks
  Percentage of patients with good or moderate response according the EULAR response criteria
Minimal disease activity (DAS28-CRP<2.9) | 24 weeks
  Percentage of patients with minimal disease activity (DAS28-CRP<2.9)
Non-responders | 24 weeks
  Percentage of patients with no response according to EULAR response criteria
Number of adverse events | 24 weeks
  The number of adverse events
Severity of adverse events | 24 weeks
  Severity of adverse events
Cumulative dose co-medication | 24 weeks
  Cumulative dose of co-medication
Times co-medication is used | 24 weeks
  Number of times co-medication is used
Cumulative dose of rescue medication | 24 weeks
  Cumulative dose of rescue medication
Times rescue medication is used | 24 weeks
  Number of times co-medication is used

CONTACTS AND LOCATIONS:
Overall Officials: Gertjan Wolbink, PhD, Principal Investigator — Reade Rheumatology Research Institute; Alfons A Den Broerder, PhD, Principal Investigator — Sint Maartenskliniek
Locations (2):
- Netherlands (2):
  - Sint Maartenskliniek, Ubbergen, Gelderland
  - Reade Rheumatology Research Institute, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: Yes
To avoid duplication of research, the gathered data will be shared once all desirable data analysis have been performed and the results are published
Supporting Information: Study Protocol, SAP
Time Frame: Six months after the study is published the data will be shared
Access Criteria: Researchers with demonstrable interest in autoimmunity, biologicals, or therapeutic drug monitoring (TDM) can contact the investigators of the trial if they are interested in gaining access to the data. Depending on their research objectives the data will be shared

REFERENCES:
- [Background] Cantini F, Niccoli L, Nannini C, Cassara E, Kaloudi O, Giulio Favalli E, Becciolini A, Benucci M, Gobbi FL, Guiducci S, Foti R, Mosca M, Goletti D. Second-line biologic therapy optimization in rheumatoid arthritis, psoriatic arthritis, and ankylosing spondylitis. Semin Arthritis Rheum. 2017 Oct;47(2):183-192. doi: 10.1016/j.semarthrit.2017.03.008. Epub 2017 Mar 22. PMID 28413099
- [Background] Hyrich KL, Lunt M, Watson KD, Symmons DP, Silman AJ; British Society for Rheumatology Biologics Register. Outcomes after switching from one anti-tumor necrosis factor alpha agent to a second anti-tumor necrosis factor alpha agent in patients with rheumatoid arthritis: results from a large UK national cohort study. Arthritis Rheum. 2007 Jan;56(1):13-20. doi: 10.1002/art.22331. PMID 17195186
- [Background] Jamnitski A, Bartelds GM, Nurmohamed MT, van Schouwenburg PA, van Schaardenburg D, Stapel SO, Dijkmans BA, Aarden L, Wolbink GJ. The presence or absence of antibodies to infliximab or adalimumab determines the outcome of switching to etanercept. Ann Rheum Dis. 2011 Feb;70(2):284-8. doi: 10.1136/ard.2010.135111. Epub 2010 Nov 10. PMID 21068090
- [Background] L' Ami MJ, Ruwaard J, Krieckaert C, Nurmohamed MT, van Vollenhoven RF, Rispens T, Wolbink GJ. Serum drug concentrations to optimize switching from adalimumab to etanercept in rheumatoid arthritis. Scand J Rheumatol. 2019 Jul;48(4):266-270. doi: 10.1080/03009742.2019.1577915. Epub 2019 Apr 23. PMID 31012365